CLINICAL TRIAL: NCT05230836
Title: Effectiveness and Safety of Electrical Stimulation With Alternating High-frequency Currents (30-50 Kilohertz) on the Sensorimotor System in Healthy Volunteer Subjects
Brief Title: HFAC Stimulation (30-50 Kilohertz) in Healthy Volunteers (High Frequency Alternating Current Stimulation)
Acronym: HFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: neuromodest-gifto; 2021-006548-28 (EudraCT Number); MCIN/10.13039/501100011033 (Other: Ministery of science and innovation of Spain)
Record Dates: First submitted 2022-01-14; First posted 2022-02-09 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Healthy; Nerve Block; Pain
Keywords: high-frequency alternating current stimulation; Nerve block; Pain; Strength; Median nerve
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Four interventions will be performed in randomized order: Group A: 30 kHz HFAC, group B: 40 kHz HFAC, group C: 50 kHz HFAC and group D: simulated electrical stimulation.
  kHz (kilohertz)
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants and evaluator shall be performed using the same equipment, electrodes, cables, and placement for the actual or placebo treatments. In addition, the participants and the evaluator will not have a view of the equipment screen. Blinding of the outcome assessor will be performed using different team members for randomization of the interventions (Investigator 1), intervention (Investigator 2), evaluation (Investigator 3) and statistical analysis (Investigator 4). Randomization will be kept hidden from participants and research team members in sealed envelopes and only the researcher who will deliver the intervention (researcher 2) will know the group assignment. Successful blinding of participants and evaluator will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30 kilohertz (Experimental): Alternating current stimulation at 30 kilohertz via transcutaneous, 15 minutes each intervention with a maximum intensity of 400 milliamperes (mA).
  Interventions: Other: High-frequency alternating current stimulation
- 40 kilohertz (Experimental): Alternating current stimulation at 40 kilohertz via transcutaneous, 15 minutes each intervention with a maximum intensity of 400 milliamperes (mA).
  Interventions: Other: High-frequency alternating current stimulation
- 50 kilohertz (Experimental): Alternating current stimulation at 50 kilohertz via transcutaneous, 15 minutes each intervention with a maximum intensity of 400 milliamperes (mA).
  Interventions: Other: High-frequency alternating current stimulation
- Sham stimulation (Sham Comparator): Sham stimulation via transcutaneous, 15 minutes each intervention, following the same procedures as 30, 40 and 50kHz HFAC groups.
  Interventions: Other: Sham current stimulation

INTERVENTIONS:
Other: High-frequency alternating current stimulation — For electrical stimulation in the active groups, unmodulated alternating currents with a symmetrical rectangular waveform of 30 kHz, 40 kHz and 50 kHz will be applied. The current intensity shall be adjusted individually for each participant by increasing the current intensity until the participant reports a "strong but comfortable tingling" sensation just below the excitomotor threshold on the palmar aspect of the hand in the dermatomes innervated by the median nerve. The intensity of the current shall be adjusted every two minutes if the tingling sensation decreases. This protocol has been used in previous studies conducted by our research group
  Other Names: Neuromodest® Cibertec-Inc. CHFS 500i
  Arms: 30 kilohertz; 40 kilohertz; 50 kilohertz
Other: Sham current stimulation — Sham electrical stimulation will be performed with the same equipment and electrodes as in the active groups without the participants and the evaluator having a view of the device screen. The intensity of the current will be increased for 30 seconds until the sensory threshold ("strong but comfortable tingling sensation") is exceeded and once the threshold is reached, the intensity will be reduced to 0 mA with 30 seconds ramp down. Participants will not receive electrical current during the rest of the placebo intervention. This protocol was used in other studies with similar interventions to blind participants.
  Other Names: Neuromodest® Cibertec-Inc. CHFS 500i sham
  Arms: Sham stimulation

SUMMARY:
High-frequency alternating current (HFAC) stimulation (between 1 kilohertz (kHz) and 100 kHz) on the peripheral nerve has been shown in basic animal research to produce a rapidly reversible nerve block without nerve damage. In human studies, frequencies between 1 kHz and 30 kHz had been applied (both transcutaneously and percutaneously), showing rapidly reversible sensorimotor changes after stimulation without adverse effects. However, the effect of currents with a frequency higher than 30 kHz, which has been shown to be more effective in eliciting nerve block in primates, has not been investigated in humans.

The main objective of this study is to investigate the safety of the intervention and the effect in healthy volunteers of transcutaneous application of alternating currents with frequencies between 30 kHz and 50 kHz on neurophysiological changes in the nerve (nerve conduction velocity and antidromic sensory action potentials (SNAPs), sensory (pain to pressure, epicritic sensitivity and thermal pain to heat) and motor (maximal isometric force) components of the median nerve.

DETAILED DESCRIPTION:
Electrical stimulation with high-frequency alternating currents (between 1 kHz and 100 kHz) on the peripheral nerve has shown, in basic research with animals, that it produces a rapidly reversible nerve block without causing damage to the nerve. In humans, studies have been carried out with frequencies between 1 kHz and 30 kHz applied both transcutaneously and percutaneously, showing rapidly reversible sensorimotor changes after stimulation and without causing adverse effects. However, the effect of currents with a frequency greater than 30 kHz has not been investigated in humans, which has been shown to be more effective in causing nerve block in primates.

The main objective of this study is to investigate the safety of the intervention and the effect in healthy volunteers of the transcutaneous application of alternating currents with frequencies between 30 kHz and 50 kHz on neurophysiological changes in the nerve (nerve conduction velocity and antidromic sensory compound action potentials (PACSA), the sensitive component (pressure pain, epicritic sensitivity and thermal pain to heat) and motor (maximum force) of the median nerve.

A randomized, double-blind, placebo-controlled crossover clinical trial has been designed. The participants will be healthy volunteers between 18 and 40 years old recruited from the students and staff of the Faculty of Physiotherapy and Nursing of the University of Castilla-La Mancha. Four interventions will be performed randomizing the order: Group A: 30 kHz, group B: 40 kHz, group C: 50 kHz and group D: sham electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer participants.
* Ability to perform all clinical tests and understand the study protocol, as well as obtain informed consent.
* Tolerance to the application of electrotherapy.

Exclusion Criteria:

* Having been treated with an electric current similar to the one applied prior to the intervention.
* Neurological pathology of peripheral or central origin.
* Altered sensitivity in the area of application of the intervention.
* No compromise of continuity.
* History of neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb.
* Diabetes.
* History of cancer.
* Cardiovascular, metabolic or immunological diseases.
* Presence of pacemaker or any other implanted electrical device.
* Taking medication during the study and in the 7 days prior to the study.
* Consumption of narcotic substances during the study and in the 7 days prior to the study.
* Presence of tattoos or any other external agent introduced in the area of treatment and treatment and assessment area (hand).
* Pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  It will be assessed as an indirect measure of the blockade of the Aδ sensory fibers of the median nerve. Once the applicator is placed perpendicular to the skin, over an uncomfortable spot on the palmar aspect of the non-dominant hand, the pressure shall be increased at a rate of approximately 5 N/s. Three measurements shall be taken with an interval between measurements of 15 seconds, the average of the three measurements shall be taken as the pressure pain threshold.

SECONDARY OUTCOMES:
Compound antidromic sensitive nerve action potentials | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  It will be assessed as a direct measure of blockade of the large diameter sensory fibers Aα and Aβ over the non-dominant hand. Two recording electrodes (model Repusi-Gwc-1.5r reusable conductive ring electromyography electrodes) shall be used and placed on the index finger, the anode over the metacarpophalangeal joint and the cathode over the distal interphalangeal joint. The ground electrode shall be placed over the styloid process of the radius. The location of the median nerve in the forearm is then identified by transcutaneous bipolar stimulation. To evoke the action potential, supramaximal stimuli will be applied using a pulse width of 1000µs at a frequency of 1 Hz. The average of a train of 10 pulses will be collected for subsequent analysis.
Maximal isometric pinch strength | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  It will be assessed as an indirect measure of the blockade of the motor fibers (Aα motor neurons) of the median nerve. Assessment of palmar pincer isometric peak force of the non-dominant hand (distal phalanx of the second and third finger with the distal phalanx of the first finger) shall be performed with a pincer dynamometer (Pinch meter P200 Biometric LTD). Three measurements of the peak isometric pincer force in Kg/f shall be recorded and the average of the three measurements shall be taken as the peak force value. The subject will hold the force for at least 3 seconds and it will be performed progressively until the maximum peak is reached, with at least 15 seconds of recovery between measurements. This measurement has shown excellent validity and reliability for measuring strength in median nerve blocks and neurological pathologies.
Two points discrimination threshold | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  This will be assessed as an indirect measure of the blockage of the Aβ sensory fibers of the median nerve. Two-point tactile discrimination between two points will be carried out on the anterior face of the distal phalanx of the third finger with an esthesiometer (Baseline®). This evaluation will be carried out according to the protocol described by Sang W. et al (2017), instructing the subject to report when they perceive a point or two. The protocol begins with a descending trial with the esthesiometer initially set at a distance of 10 mm and decreasing by 1 mm until the participant reports perceiving a single point. When that happens, several stimuli around that threshold will be given randomly, including stimuli with a single tip. If the subject correctly identifies two of three stimuli while not at a shorter distance, that will be considered their final discrimination threshold.
Heat pain threshold | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  It will be assessed as an indirect measure of the blockade of the type C amyelinic sensory fibers of the median nerve. Hot thermal stimuli will be applied over the thenar eminence in the palmar aspect of the non-dominant hand (dermatome innervated by the median nerve), using a 9 cm2 thermoelectric cell (TSA 2. Medoc, Israel). Three temperature ramp-up measurements will be performed with a time between tests of 30 seconds. The thermal pain threshold to heat shall be determined by the limit method and the mean value of the 3 measurements shall be taken as the threshold value. The starting temperature shall be 32°C and the rate of ascent shall be 1°C/s, with a rate of descent of 8,5°C/s. Subjects shall be instructed to press the device with the contralateral hand when the warm thermal sensation becomes painful and the temperature of the applicator shall automatically decrease. For safety reasons, 50°C shall be set as the cut-off temperature.
Skin temperature | Baseline, during intervention at 10 minutes, post immediate at 15 minutes and 15 minutes post intervention.
  A doppler temperature and perfusion monitor (Moor Instruments model DRT4) with a recording sensor placed on the palmar side over the head of the third metacarpal will be used to record skin temperature of the non-dominant hand. An external analog thermometer shall be used to record the ambient temperature.
Adverse effects and subjective current sensations | Post immediate at 15 minutes and 24 hours after the intervention
  In order to assess the adverse effects and the subjective perception of the participants, a standardized questionnaire was developed. In this questionnaire, ten items have been established with response options (YES/NO) in relation to heat, cold, sweating, tingling, pain (burning/punching/electrical, superficial/deep), numbness, numbness, stiffness/shrinking, heaviness and/or weakness, together with the area in which they are perceived and an open item in which other effects or sensations that the participant has perceived will be collected. The unpleasantness of the intervention will also be assessed using a 10 cm visual analog scale where 0 corresponds to "not at all unpleasant" and 10 to "as unpleasant as you could receive".
Outcome and participant blinding assessment | Post immediate at 15 minutes each intervention.
  Immediately after stimulation intervention (15 min) (30, 40, 50 kHz and sham) the success of blinding will be assessed through five response options: "What type of intervention do you think you have received?" I strongly believe I have received an experimental treatment/ I slightly believe I have received an experimental treatment/ I strongly believe I have received a placebo/ I slightly believe I have received a placebo/ don't know or no answer.

OTHER OUTCOMES:
Demographic characteristics | Pre intervention (baseline 0min)
  Demographic characteristics as age in years, gender, dominant upper limb, weight in kilograms, height in metres and body mass index in kg/m2 will be recorded. It shall also be recorded that the subject does not show any exclusion criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Principal Investigator — University of Castilla-La Mancha; Julio Gómez-Soriano, PhD, Study Director — University of Castilla-La Mancha; Diego Serrano-Muñoz, PhD, Study Chair — University of Castilla-La Mancha; Juan José Fernández-Pérez, PhD student, Study Chair — University of Castilla-La Mancha
Locations (1):
- Castilla-La Mancha University, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, figures, images and appendix)
Supporting Information: Study Protocol, SAP
Time Frame: 1 month following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent ethical committee identified for this purpose.
  This data will be shared only for individual participant data meta-analysis. The proposal should be directed to juan.avendano@uclm.es. The investigator will need to sign a data access agreement. Data will be available for 5 years.

REFERENCES:
- [Background] Megia Garcia A, Serrano-Munoz D, Bravo-Esteban E, Ando Lafuente S, Avendano-Coy J, Gomez-Soriano J. [Analgesic effects of transcutaneous electrical nerve stimulation (TENS) in patients with fibromyalgia: A systematic review]. Aten Primaria. 2019 Aug-Sep;51(7):406-415. doi: 10.1016/j.aprim.2018.03.010. Epub 2018 Jul 17. Spanish. PMID 30029964
- [Background] Serrano-Munoz D, Avendano-Coy J, Simon-Martinez C, Taylor J, Gomez-Soriano J. 20-kHz alternating current stimulation: effects on motor and somatosensory thresholds. J Neuroeng Rehabil. 2020 Feb 19;17(1):22. doi: 10.1186/s12984-020-00661-x. PMID 32075666
- [Background] Serrano-Munoz D, Avendano-Coy J, Simon-Martinez C, Taylor J, Gomez-Soriano J. Effect of high-frequency alternating current transcutaneous stimulation over muscle strength: a controlled pilot study. J Neuroeng Rehabil. 2018 Nov 12;15(1):103. doi: 10.1186/s12984-018-0443-2. PMID 30419966
- [Derived] Fernandez-Perez JJ, Serrano-Munoz D, Gomez-Soriano J, Alvarez DM, Avendano-Coy J. Selective nociceptive modulation using a novel prototype of transcutaneous kilohertz high-frequency alternating current stimulation: a crossover double-blind randomized sham-controlled trial. J Neuroeng Rehabil. 2024 Nov 15;21(1):203. doi: 10.1186/s12984-024-01503-w. PMID 39548560